CLINICAL TRIAL: NCT00265148
Title: Effects of Avandia on Cognition and Cerebral Glucose Utilisation in Subjects With Mild to Moderate Alzheimer's Disease (AD).
Brief Title: Brain Imaging Study Of Rosiglitazone Efficacy And Safety In Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRL-49653/461; 2005-005089-34 (EudraCT Number)
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Alzheimer's Disease
Keywords: rosiglitazone; cognition; cerebral glucose metabolism; positron emission tomography (PET); Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosiglitazone (Experimental): 4 mg once a day for 1 month increasing to 8 mg once a day (Extended Released Tablets)
  Interventions: Drug: Rosiglitazone
- Placebo (Other): Placebo dummy to match
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rosiglitazone — Extended Release Tablets
  Arms: Rosiglitazone
Other: Placebo — Placebo dummy to match
  Arms: Placebo

SUMMARY:
This is a placebo-controlled study evaluating the effects of rosiglitazone on functional brain activity and cognition in patients with mild to moderate Alzheimer's Disease (AD).

ELIGIBILITY:
Inclusion criteria:

* Is male, or if female meets one or more of the following criteria:
* Post-menopausal females defined as menopause is defined as>6months without menstrual period with an appropriate clinical profile, e.g. age appropriate, history of vasomotor symptoms. However if indicated this should be confirmed by oestradiol and FSH levels consistent with menopause (according to local laboratory ranges). Women who are on HRT treatment, and have not been confirmed as post-menopausal should be advised to use contraception.(See Appendix 4)Pre-menopausal females with a documented (medical report verification) hysterectomy and/or bilateral oophorectomy only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Meets the National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for Alzheimer's disease, regardless of date of diagnosis relative to study entry date. (See Appendix 5) Has an Alzheimer's disease status of mild to moderate, as classified by a Mini Mental State Examination (MMSE) score of 16-26 inclusive at screening.

Is aged >/= 50 to </= 85 years Prior and current use of medication corresponds with criteria listed in Appendix 3.

* Has the ability to comply with requirements of cognitive and other testing.
* Has a permanent caregiver who is willing to attend all visits, oversee the subject's compliance with protocol-specified procedures and study medication, and report on subject's status. (Subjects living alone or in a nursing home are not eligible).
* Has provided full written informed consent prior to the performance of any protocol-specified procedure; or if unable to provide informed consent due to cognitive status, provision of informed consent by cognitively intact legally acceptable representative (Where this is in accordance with local laws, regulations and ethics committee policy.) Caregiver has provided full written informed consent prior to the performance of any protocol-specified procedure.

Exclusion criteria:

* Is unsuitable for MRI scanning as assessed by local pre-MRI questionnaire (GSK to review.)
* Has a history of or suffers from claustrophobia.
* Is unable to lie comfortably on a bed inside a PET camera with their head in the field of view for at least 60 minutes as assessed by physical examination and medical history (e.g. back pain, arthritis).
* Has a history or presence of other neurological or other medical conditions that may influence the outcome or analysis of the PET scan results. Examples of such conditions include, but are not limited to stroke, traumatic brain injury, epilepsy or space occupying lesions.
* History of Type I or Type II diabetes mellitus.
* Fasting plasma glucose level>126mg/dL (>7.0mmol/L) or HbA1c>6.2%.
* History or clinical/laboratory evidence of moderate congestive heart failure defined by the New York Heart Association criteria (class I-IV)(See Appendix 6).

Ejection fraction</=40% determined by echocardiogram, or any other abnormality on echocardiography which in the view of the investigator required further investigation or intervention, or significant abnormalities on screening ECG (in accordance with the definitions below). Significant ECG abnormalities for the purposes of this study. Detection of any of the following abnormalities renders the subject ineligible for the study: 1. ECG heart rate <50 and >100 bpm 2. Any previously unrecognised sustained or paroxysmal arrhythmia requiring further intervention e.g. anticoagulation, cardioversion, anti-arrhythmic agent, further investigation etc. 3. PR interval >0.3 s, 2nd or 3rd degree heart block, symptomatic bifascicular block, trifascicular block. 4. Multifocal ventricular ectopy. 5. Ventricular bigemini or couplets, triplets etc. ECG abnormalities permitted at entry to this study. A subject will not be rendered ineligible by the presence of any of the following abnormalities: 1. AF with a heart rate <=90 in subjects receiving appropriate anti-platelet or anticoagulant therapy. 2. 1st degree heart block (PR<=0.3 s). 3. Subjects with a paced rhythm (further information required if subject has an implantable Cardiac Defibrillator). 4. Atrial ectopic beats. 5. Unifocal ventricular ectopic beats. 6. Left or right bundle branch block. 7. Asymptomatice bifascicular block. 8. Left ventricular hypertrophy. 9. Q waves present suggesting previous MI. 10. Repolarisation abnormalities History of new cardiovascular event within the last 6 months (i.e. intervention, percutaneous coronary intervention, vascular surgery, acute coronary syndrome [non Q-wave myocardial infarction, Q-wave myocardial infarction, unstable angina) or significant arrhythmia; or major intervention (e.g. cardiac surgery or angiography plus stenting) scheduled.

* History or clinical laboratory evidence of cerebrovascular disease (stroke, transient ischaemic attack, haemorrhage), or diagnosis of possible, probable or definite vascular dementia in accordance with National Institute of Neurological Disorders and Stroke, and Association Internationale pour la Recherche et l'Enseignement en Neurosciences (NINDS-AIREN) criteria (See Appendix 8).
* History or evidence of any other CNS disorder that could be interpreted as a cause of dementia: e.g. structural abnormality, epilepsy, infectious or inflammatory/demyelinating CNS conditions, Parkinson's disease.

Significant peripheral oedema at the time of screening as assessed by Clinical Evaluation of Oedema and/or Signs of Congestive Heart Failure (Appendix 14)

* History of major psychiatric illness such as schizophrenia or bipolar affective disorder, or current depression (score on Hospital Anxiety and Depression Scale (HADS) depression questions >7, See Appendix 9).

Systolic blood pressure >165 mmHg or diastolic blood pressure >95 mmHG whilst receiving optimal antihypertensive therapy according to local practice.

Clinically significant anaemia (i.e.haemoglobin <11g/dL for males or <10 g/dL for females) or presence of haemoglobinopathies which would prevent accurate assessment of HbA1c.

Renal dysfunction, defined as creatinine clearance <30 ml/min (calculated from serum creatinine using the Cockcroft-Gault formula, See Appendix 10).

ALT, AST, total bilirubin, or alkaline phosphatase >2.5 times the upper limit of normal laboratory range, or history of severe hepatobiliary disease (e.g. hepatitis B or C, or cirrhosis (Childs-Pugh classes B/C)) without enzyme elevation.

* Fasting triglycerides >12mmol/L Abnormal/positive result within the past 12 months or at screening for any of the following tests: vitamin B12 (</=200pg/mL), syphilis serology, thyroid stimulating hormone.
* History or presence of gastro-intestinal, hepatic or renal disease or other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.

any clinically relevant abnormality, medical or psychiatric condition, which, in the opinion of the investigator, makes the subject unsuitable for inclusion in the study.

* Has donated >/= ml of blood within the past 2 months. Use of any other investigational agent within 30 days or 5 half-lives (whichever is longer) prior to the screening visit.

History of alcohol abuse, or of drug abuse within the past 6 months (or has tested positive for drugs of abuse at screening).

Subject is unable (with assistance, if appropriate) to take study medication as prescribed throughout the study.

* History of non-compliance with prescribed medication, or risk of non-compliance with study medication or procedures.

Subject is an immediate family member or employee of the participating investigator or of any of the participating site staff.

Shows any neurological abnormality by MRI, which in the opinion of the Principal Investigator would introduce additional risk factors, study procedures or effect endpoint data. MRI scanning will only be conducted on subjects who satisfy all other eligibility criteria.

* History of bone marrow transplant Exhibits screening/baseline results not consistent with AD e.g. radiological findings, or results on cognitive tests.

Use of tacrine within 30 days prior to the screening visit.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-05-18 (Actual); Primary Completion 2008-07-10 (Actual); Study Completion 2008-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (9):
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Belmont, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Durham, North Carolina
- GSK Investigational Site, Montreal, Quebec, Canada
- United Kingdom (4):
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Swindon
  - GSK Investigational Site, West End, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Tzimopoulou S, Cunningham VJ, Nichols TE, Searle G, Bird NP, Mistry P, Dixon IJ, Hallett WA, Whitcher B, Brown AP, Zvartau-Hind M, Lotay N, Lai RY, Castiglia M, Jeter B, Matthews JC, Chen K, Bandy D, Reiman EM, Gold M, Rabiner EA, Matthews PM. A multi-center randomized proof-of-concept clinical trial applying [(1)(8)F]FDG-PET for evaluation of metabolic therapy with rosiglitazone XR in mild to moderate Alzheimer's disease. J Alzheimers Dis. 2010;22(4):1241-56. doi: 10.3233/JAD-2010-100939. PMID 20930300
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: BRL-49653/461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: BRL-49653/461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: BRL-49653/461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: BRL-49653/461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: BRL-49653/461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: BRL-49653/461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: BRL-49653/461 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 18 May 2004 to 10 July 2008 at centers across Canada, the United States (US), and the United Kingdom (UK). A total of 80 participants with mild to moderate Alzheimer's disease were planned to be enrolled.
Pre-assignment Details: A total of 135 participants were screened of which 80 participants were randomized, during which they received oral Rosiglitazone-extended (RSG-XR) release 4 milligrams (mg) once daily. Intent- to-treat (ITT) population included 78 participants who had more than or equal to 1 efficacy, pharmacokinetic, pharmacodynamics, or genetic assessment.
Groups:
- Placebo: Eligible participants received unit oral dose of visually matching Placebo 4 milligrams (mg) for one month. Participants received escalated dose of 8 mg matching placebo for next 12 months and were followed-up to 30 days.
- Rosiglitazone: Eligibale participants received unit oral Rosiglitazone extended release (RSG XR) 4 mg for one month with or without food. Participants received escalated dose of rosiglitazone-XR for next 12 months and were followed-up to 30 days.
Period: Overall Study
Arm/Group | Placebo | Rosiglitazone
Started | 40 | 40
Completed | 31 | 31
Not Completed | 9 | 9
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Increasing frailty | 0 | 1
Not completed — Subject chose to change of the dose | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants from all subjects population who had at least one or more than one post-baseline pharmacodynamic (PD) or biomarker, efficacy, or pharmacogenetic (PGx) assessment.
Groups:
- Rosiglitazone: Eligible participants received unit oral rosiglitazone extended release (RSG XR) 4 mg for one month with or without food. Participants received escalated dose of rosiglitazone-XR for next 12 months and were followed-up to 30 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rosiglitazone | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (9.28) | 72.5 (9.60) | 71.4 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 20 | 22 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American hispanic | 1 | 1 | 2
  Black | 1 | 0 | 1
  White/Caucasian | 37 | 37 | 74
  Other Caucasiann/ Japanese | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Day 1) in Global and Regional Indices of Cerebral Metabolic Rate of Glucose (CMRglu) at Month 12
Description: Global CMRGlu index was related to grey matter of brain. Regional CMRGlu index was related to assessment of different regions of brain namely posterior cingulate gyrus, frontal lobe, parietal lobe, posterior temporal lobe, cerebellum, and medial temporal lobe. Evaluation of medial temporal lobe CMRGlu included assessment of medial anterior temporal lobe, paraHippocampal Ambiens gyrus, amygdala, and hippocampus. The regional CMRGlu index is directly proportional to the true metabolic rate of glucose. Baseline was defined as Day 1 of the 12 months treatment period. Change from Baseline is the value at indicated time point minus the Baseline value. Data has been presented for arithmetic mean; however, statistical analysis has been presented for adjusted or least square (LS) mean.
Time Frame: Baseline (Day 1) and Month 12
Population: Intent-to-treat (ITT) population included all participants from all subjects population who had at least one or more than one post-baseline pharmacodynamic (PD) or biomarker, efficacy, or pharmacogenetic (PGx) assessment. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Milligrams per cubic centimeter(mg/cm^3)
Groups:
- Placebo: Eligible participants received unit oral dose of visually matching Placebo 4 mg for one month. Participants received escalated dose of 8 mg matching placebo for next 12 months and were followed-up to 30 days.
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Milligrams per cubic centimeter(mg/cm^3)
  Grey matter: number analyzed (Participants) | 25 | 27
  Grey matter | -0.2793 (0.48541) | -0.0887 (0.34985)
  Posterior cingulate gyrus: number analyzed (Participants) | 25 | 27
  Posterior cingulate gyrus | -0.3143 (0.57567) | -0.0786 (0.36019)
  Frontal lobe: number analyzed (Participants) | 25 | 27
  Frontal lobe | -0.3087 (0.55631) | -0.1131 (0.36876)
  Parietal lobe: number analyzed (Participants) | 25 | 27
  Parietal lobe | -0.3081 (0.50596) | -0.1175 (0.33335)
  Posterior temporal lobe: number analyzed (Participants) | 25 | 27
  Posterior temporal lobe | -0.2771 (0.40458) | -0.1122 (0.32346)
  Cerebellum: number analyzed (Participants) | 22 | 25
  Cerebellum | -0.2523 (0.46730) | -0.0248 (0.38874)
  Medial temporal lobe: number analyzed (Participants) | 25 | 27
  Medial temporal lobe | -0.1950 (0.33360) | -0.0349 (0.32429)
Statistical Analysis 1: Comparison: Placebo vs Rosiglitazone; For Grey matter; Test type: Superiority or Other; p = 0.1695, Mixed model for repeated measures; Mean Difference (Net) = 0.1334, 95% CI 2-sided [-0.0583 to 0.3251]
Statistical Analysis 2: Comparison: Placebo vs Rosiglitazone; For posterior cingulate Gyrus; Test type: Superiority or Other; p = 0.1057, Mixed model for repeated measures; Mean Difference (Net) = 0.1750, 95% CI 2-sided [-0.0380 to 0.3880]
Statistical Analysis 3: Comparison: Placebo vs Rosiglitazone; For Frontal lobe; Test type: Superiority or Other; p = 0.1833, Mixed model for repeated measures; Mean Difference (Net) = 0.1426, 95% CI 2-sided [-0.0691 to 0.3543]
Statistical Analysis 4: Comparison: Placebo vs Rosiglitazone; For parietal lobe; Test type: Superiority or Other; p = 0.1644, Mixed model for repeated measures; Mean Difference (Net) = 0.1366, 95% CI 2-sided [-0.0574 to 0.3307]
Statistical Analysis 5: Comparison: Placebo vs Rosiglitazone; For Posterior temporal lobe; Test type: Superiority or Other; p = 0.1509, Mixed model for repeated measures; Mean Difference (Net) = 0.1259, 95% CI 2-sided [-0.0471 to 0.2989]
Statistical Analysis 6: Comparison: Placebo vs Rosiglitazone; For cerebellum; Test type: Superiority or Other; p = 0.2041, Mixed model for repeated measures; Mean Difference (Net) = 0.1339, 95% CI 2-sided [-0.0747 to 0.3424]
Statistical Analysis 7: Comparison: Placebo vs Rosiglitazone; For medial temporal lobe; Test type: Superiority or Other; p = 0.1445, Mixed model for repeated measures; Mean Difference (Net) = 0.1094, 95% CI 2-sided [-0.0385 to 0.2572]

2. Secondary Outcome: Change From Baseline (Day 1) in CMRGlu Indices at Months 1 and 6
Description: Global CMRGlu index was related to grey matter of brain. Baseline measurement was performed on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1), Months 1, and 6
Population: ITT population. Only those participants available at the time of assessment were analyzed
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
mg/cm^3
  Month 1: number analyzed (Participants) | 33 | 37
  Month 1 | -0.1049 (0.39301) | 0.0475 (0.46904)
  Month 6: number analyzed (Participants) | 30 | 33
  Month 6 | -0.1556 (0.36397) | -0.0269 (0.35311)
Statistical Analysis 1: Comparison: Placebo vs Rosiglitazone; At Month 1; Test type: Superiority or Other; p = 0.2251, Mixed model for repeated measures; Mean Difference (Net) = 0.1211, 95% CI 2-sided [-0.0763 to 0.3185]
Statistical Analysis 2: Comparison: Placebo vs Rosiglitazone; For Month 6; Test type: Superiority or Other; p = 0.2497, Mixed model for repeated measures; Mean Difference (Net) = 0.0893, 95% CI 2-sided [-0.0643 to 0.2430]

3. Secondary Outcome: Change From Baseline (Day 1) in Delayed Free Recall Words at Months 1, 6, and 12 by Buschke Selective Reminding (BSR) Test
Description: The BSR test included evaluating short-term memory of a participant to remember a list of unrelated words, to learn the words over 8 trials and to remember these words over 8 trials, and to remember these words during a 20 minute delay. The number of words recalled in delayed free recalls were analyzed. Other parameters analyzed included number recalled Trial 1 immediate, number recalled Trial 8 immediate, total number for all 8 immediate trials, and total number of uncued words recalled. Higher number of words recalled indicated better short term memory and positive treatment differences in these number of words recalled were indicative of superiority of drug over placebo. Baseline measurement was performed on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value. Statistical analysis is presented for difference of means.
Time Frame: Baseline (Day 1), and Months 1, 6, and 12
Population: ITT population. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Number of words recalled
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Number of words recalled
  Delayed free recall, Month 1: number analyzed (Participants) | 32 | 34
  Delayed free recall, Month 1 | 0.1 (1.72) | 0.2 (1.23)
  Delayed free recall, Month 6: number analyzed (Participants) | 27 | 31
  Delayed free recall, Month 6 | -0.1 (1.56) | 0.0 (1.21)
  Delayed free recall, Month 12: number analyzed (Participants) | 25 | 26
  Delayed free recall, Month 12 | -0.4 (1.32) | -0.4 (1.53)
  Trial 1 immediate, Month 1: number analyzed (Participants) | 32 | 34
  Trial 1 immediate, Month 1 | 0.2 (1.30) | -0.1 (1.13)
  Trial 1 immediate, Month 6: number analyzed (Participants) | 27 | 31
  Trial 1 immediate, Month 6 | -0.2 (1.69) | -0.1 (1.42)
  Trial 1 immediate, Month 12: number analyzed (Participants) | 25 | 26
  Trial 1 immediate, Month 12 | -0.6 (1.32) | -0.5 (1.27)
  Trial 8 immediate, Month 1: number analyzed (Participants) | 32 | 34
  Trial 8 immediate, Month 1 | -0.2 (1.82) | 0.0 (1.45)
  Trial 8 immediate, Month 6: number analyzed (Participants) | 27 | 31
  Trial 8 immediate, Month 6 | -0.3 (1.29) | -0.2 (1.21)
  Trial 8 immediate, Month 12: number analyzed (Participants) | 25 | 26
  Trial 8 immediate, Month 12 | -0.9 (1.32) | -0.2 (1.03)
  For all 8 immediate trial, Month 1: number analyzed (Participants) | 32 | 34
  For all 8 immediate trial, Month 1 | -1.4 (7.27) | 0.9 (5.51)
  For all 8 immediate trial, Month 6: number analyzed (Participants) | 27 | 31
  For all 8 immediate trial, Month 6 | -3.0 (7.31) | 0.4 (5.85)
  For all 8 immediate trial, Month 12: number analyzed (Participants) | 25 | 26
  For all 8 immediate trial, Month 12 | -5.8 (7.95) | -0.9 (5.27)
  Uncued words recalled, Month 1: number analyzed (Participants) | 32 | 34
  Uncued words recalled, Month 1 | -1.7 (8.56) | 0.9 (5.43)
  Uncued words recalled, Month 6: number analyzed (Participants) | 27 | 31
  Uncued words recalled, Month 6 | -3.2 (7.92) | 0.9 (7.55)
  Uncued words recalled, Month 12: number analyzed (Participants) | 25 | 26
  Uncued words recalled, Month 12 | -7.0 (9.91) | -2.0 (8.59)
Statistical Analysis 1: Comparison: Placebo vs Rosiglitazone; For BSR test , Month 1; Test type: Superiority or Other; p = 0.7618, Repeated measure mixed model; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.59 to 0.80]
Statistical Analysis 2: Comparison: Placebo vs Rosiglitazone; For BSR test, Month 6; Test type: Superiority or Other; p = 0.8350, Repeated measure mixed model; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.53 to 0.66]
Statistical Analysis 3: Comparison: Placebo vs Rosiglitazone; For BSR test, Month 12; Test type: Superiority or Other; p = 0.6735, Repeated measure mixed model; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.78 to 0.51]

4. Secondary Outcome: Change From Baseline (Day 1) in Delayed Free Recall Items Over Period by Stroop Colour Word Interference (SCWI) at Months 1, 6 and 12
Description: It is a measure of change from Baseline (Day 1) in clinical scale of AD status. A 3-card version test includes all card containing 50 items each. Participants were asked to complete all items and time in seconds was recorded. Participants first read color words printed in black, then named the printed color of the colored patches, and finally named the printed color of the colored words. The word condition was used to verify that participants were able to read colored words and time to perform color condition was considered as ' control'. The dependent variable was the time to complete the interference condition and the test could have presented in pencil and paper or on screen, both the ways. Change from Baseline is the value at indicated time point minus the Baseline value. Statistical analysis is presented for difference of means.
Time Frame: Baseline (Day 1), Months1, 6, and 12
Population: ITT population. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Milliseconds
  Month 1: number analyzed (Participants) | 38 | 39
  Month 1 | -0.0 (0.88) | -0.4 (1.33)
  Month 6: number analyzed (Participants) | 33 | 35
  Month 6 | 0.1 (0.97) | -0.2 (1.06)
  Month 12: number analyzed (Participants) | 29 | 30
  Month 12 | 0.5 (1.09) | -0.3 (1.78)
Statistical Analysis 1: Comparison: Placebo vs Rosiglitazone; For Month 1; Test type: Superiority or Other; p = 0.7045, Repetaed measure mixed model; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.44 to 0.30]
Statistical Analysis 2: Comparison: Placebo vs Rosiglitazone; For Month 6; Test type: Superiority or Other; p = 0.8181, Repeated measure mixed model; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.40 to 0.32]
Statistical Analysis 3: Comparison: Placebo vs Rosiglitazone; AT Month 12; Test type: Superiority or Other; p = 0.7688, Repeated measure mixed model; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.71 to 0.53]
Statistical Analysis 4: Comparison: Placebo vs Rosiglitazone; Overall; Test type: Superiority or Other; p = 0.6810, Repeated measure mixed model; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.40 to 0.26]

5. Secondary Outcome: Change From Baseline (Day 1) in Simplified Spatial Paired Associate Learning (SSPAL) Response Over Period
Description: Change from Baseline = value at the indicated time point minus the Baseline(Day1) value. SSPAL is a cognitive test that involves object-location memory and learning. It is used to examine cognitive deficits in AD. Participants were asked to sit 50 cm away from screen and different pictures (target and distracter) were shown on a monitor. Responses were acquired from response box. Participants were informed by visual feedback whether the response was correct or incorrect and the accuracy was collected automatically. SSPAL responses were captured as new accuracy and global accuracy. New accuracy was defined as proportion of accurate responses per participant for recall of any new item (picture). Global accuracy was defined as proportion of accurate responses per participant for recall of all new items and their displayed locations (i.e. right or left position on the screen). The possible range for new and global accuracy is 0(worst) to 1(best). Higher values indicate better performance.
Time Frame: Baseline (Day 1), Months 1, 6, and 12
Population: ITT population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of accurate responses
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Proportion of accurate responses
  Global accuracy, Month 1: number analyzed (Participants) | 29 | 25
  Global accuracy, Month 1 | -0.0 (0.16) | 0.0 (0.06)
  Global accuracy, Month 6: number analyzed (Participants) | 25 | 24
  Global accuracy, Month 6 | -0.0 (0.14) | -0.0 (0.12)
  Global accuracy, Month 12: number analyzed (Participants) | 21 | 21
  Global accuracy, Month 12 | -0.0 (0.15) | 0.0 (0.12)
  New accuracy, Month 1: number analyzed (Participants) | 29 | 25
  New accuracy, Month 1 | 0.1 (0.22) | 0.0 (0.17)
  New accuracy, Month 6: number analyzed (Participants) | 25 | 24
  New accuracy, Month 6 | 0.0 (0.19) | -0.0 (0.29)
  New accuracy, Month 12: number analyzed (Participants) | 21 | 21
  New accuracy, Month 12 | -0.0 (0.22) | -0.1 (0.22)

6. Secondary Outcome: Change From Baseline (Day 1) in Accuracy by Choice Reaction Time (CRT) Test Over Period
Description: A motor reaction task was presented 4 runs of 50 trials each. In each trial, presentation of a central crosshair for 200 milliseconds (ms) was followed by display of a grey square for 800 ms. The square appeared in two of five possible positions relative to the crosshair (leftmost or rightmost). When the grey square became white, the participant was trained to press the a button. In each trial of the Simple Reaction Time Task, presentation of a central crosshair for 200 ms was followed by display of one square for 800 ms. For both simple and choice versions of the task, trial duration was 4000 ms maximum. The participant was immediately informed (by color changes of the white square) whether the response to each trial was correct or incorrect, and accuracy and reaction time (RT) are automatically calculated. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) and up to 12 months
Population: ITT population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Percent accuracy
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Percent accuracy
  Accuracy, Left, Month 1: number analyzed (Participants) | 33 | 32
  Accuracy, Left, Month 1 | -0.0 (0.04) | 0.0 (0.15)
  Accuracy, Left, Month 6: number analyzed (Participants) | 30 | 30
  Accuracy, Left, Month 6 | -0.1 (0.16) | 0.0 (0.14)
  Accuracy, Left, Month 12: number analyzed (Participants) | 28 | 25
  Accuracy, Left, Month 12 | -0.1 (0.14) | 0.0 (0.12)
  Accuracy, Right, Month 1: number analyzed (Participants) | 33 | 32
  Accuracy, Right, Month 1 | 0.0 (0.02) | 0.0 (0.15)
  Accuracy, Right, Month 6: number analyzed (Participants) | 30 | 30
  Accuracy, Right, Month 6 | -0.0 (0.02) | 0.0 (0.15)
  Accuracy, Right, Month 12: number analyzed (Participants) | 28 | 25
  Accuracy, Right, Month 12 | -0.0 (0.13) | 0.0 (0.14)

7. Secondary Outcome: Change From Baseline in Cognitive Test by Simple Reaction Time (SRT) Method Over Period
Description: A motor reaction task was presented 4 runs of 50 trials each. In each trial, presentation of a central crosshair for 200 milliseconds (ms) was followed by display of a grey square for 800 ms. The square appeared in two of five possible positions relative to the crosshair (leftmost or rightmost). When the grey square became white, the participant was trained to press the a button. In each trial of the Simple Reaction Time Task, presentation of a central crosshair for 200 ms was followed by display of one square for 800 ms. For both simple and choice versions of the task, trial duration was 4000 ms maximum. The participant was immediately informed (by color changes of the white square) whether the response to each trial was correct or incorrect, and accuracy and reaction time (RT) are automatically calculated. Baseline measurement was performed on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) and up to 12 months
Population: ITT population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Milliseconds
  Month 1: number analyzed (Participants) | 33 | 32
  Month 1 | -17.1 (161.70) | 36.5 (162.72)
  Month 6: number analyzed (Participants) | 31 | 32
  Month 6 | 37.8 (170.67) | 59.3 (158.32)
  Month 12: number analyzed (Participants) | 29 | 27
  Month 12 | 177.7 (359.91) | 76.4 (179.78)

8. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Scale (ADAS-COG) Total Score Over Period
Description: Change from Baseline is the value at indicated time point minus the Baseline value. ADAS-COG is a 13 item, 11 questionnaire assessment of range of cognitive abilities including memory, comprehension, orientation in time and place, and spontaneous speech. The scale ranges from 0 to 70, with negative changes from Baseline indicating the improvement and positive changes indicating worsening of condition. Arithmetic means are presented as raw data; however, statistical analysis is based on LS means.
Time Frame: Baseline (Day 1), and Months 1, 6, and 12
Population: ITT population. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Scores on a scale
  Month 1 | -0. (5.38) | -0.5 (4.84)
  Month 6: number analyzed (Participants) | 34 | 35
  Month 6 | 1.7 (6.73) | 3.2 (5.58)
  Month 12: number analyzed (Participants) | 31 | 31
  Month 12 | 5.7 (7.52) | 6.6 (7.80)
Statistical Analysis 1: Comparison: Placebo vs Rosiglitazone; At Month 1; Test type: Superiority or Other; p = 0.8593, Repeated measure mixed model; Mean Difference (Net) = -0.20, 95% CI 2-sided [-2.38 to 1.99]
Statistical Analysis 2: Comparison: Placebo vs Rosiglitazone; At Month 6; Test type: Superiority or Other; p = 0.3201, Repeated measure mixed model; Mean Difference (Net) = 1.44, 95% CI 2-sided [-1.43 to 4.32]
Statistical Analysis 3: Comparison: Placebo vs Rosiglitazone; At Month 12; Test type: Superiority or Other; p = 0.2627, Repeated measure mixed model; Mean Difference (Net) = 2.18, 95% CI 2-sided [-1.68 to 6.04]
Statistical Analysis 4: Comparison: Placebo vs Rosiglitazone; For overall period; Test type: Superiority or Other; p = 0.3633, Repeated measure mixed model; Mean Difference (Net) = 1.14, 95% CI 2-sided [-1.35 to 3.64]

9. Secondary Outcome: Change From Baseline in Clinician Based Impression of Change-plus (CBIC +) Score Over Period
Description: The CBIC+ assessment for global functioning consists of a 7 point rating scale of severity and change with 1 indicating marked improvement and 7 indicating marked worsening. This scale was used to analyze clinically relevant effect. This was supposed to be performed by an independent investigator who is not a part of the ongoing study. Change from Baseline is the value at indicated time point minus the Baseline value. This scale was used to decide clinical status of AD. Arithmetic means are presented as raw data; however, statistical analysis has been presented for LS means.
Time Frame: Baseline (Day 1) and Months 1, 6, and 12
Population: ITT population. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Scores on a scale
  Month 1: number analyzed (Participants) | 36 | 37
  Month 1 | 3.9 (1.08) | 3.9 (0.95)
  Month 6: number analyzed (Participants) | 34 | 35
  Month 6 | 4.7 (0.93) | 4.5 (1.22)
  Month 12: number analyzed (Participants) | 31 | 31
  Month 12 | 4.9 (1.03) | 4.8 (1.38)
Statistical Analysis 1: Comparison: Placebo vs Rosiglitazone; For overall period; Test type: Superiority or Other; p = 0.5647, Repetaed measure mixed model; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.48 to 0.26]
Statistical Analysis 2: Comparison: Placebo vs Rosiglitazone; For Month 1; Test type: Superiority or Other; p = 0.9935, Repeated measure mixed model; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.46 to 0.46]
Statistical Analysis 3: Comparison: Placebo vs Rosiglitazone; At Month 6; Test type: Superiority or Other; p = 0.3794, Repeated measure mixed model; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.72 to 0.28]
Statistical Analysis 4: Comparison: Placebo vs Rosiglitazone; At Month 12; Test type: Superiority or Other; p = 0.7357, Repeated measure mixed model; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.70 to 0.49]

10. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory Score Over Period
Description: The NPI assesses the frequency and severity of behavioral disturbances in dementia across 10 domains. The total NPI score was calculated by adding all individual domains cores. The scale ranges from 0 to 120 , 0 indicating no / least burden and 120 indicating maximum burden. A negative change from Baseline indicated improvement. Baseline measurement was performed on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1), Months 1, 6 and 12
Population: ITT population. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Scores on a scale
  Month 1: number analyzed (Participants) | 31 | 32
  Month 1 | -1.6 (6.30) | -2.6 (6.82)
  Month 6: number analyzed (Participants) | 28 | 30
  Month 6 | 2.1 (8.63) | -0.8 (11.59)
  Month 12: number analyzed (Participants) | 25 | 27
  Month 12 | 0.9 (8.39) | 1.8 (13.84)

11. Secondary Outcome: Change From Baseline in Mini-mental State Examination (MMSE) Score Over Period
Description: The MMSE consists of 11 categories of orientation, memory (recent and immediate), concentration, language, and praxis. The scale ranges from 0 to 30 with lower scores indicating greater cognitive impairment. Negative changes from Baseline indicate improvement and positive changes indicate increasing symptoms. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1), and up to Month 12
Population: ITT population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 30 | 30
Scores on a scale | -3.3 (4.09) | -2.6 (3.27)

12. Secondary Outcome: Change From Baseline in Normalized Brain Volume Over Period
Description: Normalized brain volume is a function of global changes in brain structure. Reduction in brain volume is indicative of reduction in Grey matter and thus the AD stage. The method used was structural magnetic resonance imaging (MRI). Change from Baseline is the value at indicated time point minus the Baseline value. Arithmetic means have been presented; however, statistical analysis is based upon the least square (LS) means.
Time Frame: Baseline (Day 1), Month 6 and Month 12
Population: ITT population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Cubic millimeter
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Cubic millimeter
  Month 6: number analyzed (Participants) | 28 | 33
  Month 6 | -4553.1 (43069.12) | -15995.6 (41075.95)
  Month 12: number analyzed (Participants) | 27 | 29
  Month 12 | -16599.9 (47173.85) | -13929.6 (31031.06)
Statistical Analysis 1: Comparison: Placebo vs Rosiglitazone; At Month 6; Test type: Superiority or Other; p = 0.6299, Repeated measure mixed model; Arithmetic means have been presented; however, statistical analysis is based upon the least square (LS) means; Mean Difference (Net) = -4971.6, 95% CI 2-sided [-255515.6 to 15572.4]
Statistical Analysis 2: Comparison: Placebo vs Rosiglitazone; At Month 12; Test type: Superiority or Other; p = 0.2184, Repeated measure mixed model; Mean Difference (Net) = 12223.0, 95% CI 2-sided [-7450.6 to 31896.5]

13. Secondary Outcome: Percent Change From Baseline in Brain Volume Over Period
Description: Percent volume change of brain is a function of global changes in brain structure. Reduction in brain volume is indicative of reduction in Grey matter and thus the AD stage. The method used was structural magnetic resonance imaging (MRI). Baseline value was recorded on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value. Arithmetic means have been presented; however, statistical analysis is based upon the LS means.
Time Frame: Baseline (Day 1), Month 6, and Month 12
Population: ITT population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Percent change
  Month 6: number analyzed (Participants) | 21 | 28
  Month 6 | -0.9 (0.62) | -1.4 (0.94)
  Month 12: number analyzed (Participants) | 19 | 28
  Month 12 | -2.4 (1.40) | -2.6 (1.48)
Statistical Analysis 1: Comparison: Placebo vs Rosiglitazone; For Month 6; Test type: Superiority or Other; p = 0.0129, Repeated measure mixed model; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.0 to -0.1]
Statistical Analysis 2: Comparison: Placebo vs Rosiglitazone; For Month 12; Test type: Superiority or Other; p = 0.5607, Repeated measure mixed model; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.0 to 0.6]

14. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Month 12
Description: Fasting plasma glucose are indicative of Glucose metabolism. Baseline measurement was performed on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) and Month 12
Population: ITT population. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 27 | 28
Millimoles per Liter | 0.2556 (0.99974) | -0.1750 (0.48810)

15. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin [HbA1C] at Month 12
Description: HbA1c levels are measure of glucose metabolism in body. Baseline value measurement was performed on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) and Month 12
Population: ITT population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 32 | 31
Percentage of HbA1c | 0.0625 (0.43533) | 0.3871 (0.49514)

16. Secondary Outcome: Change From Baseline in Lipid (Cholesterol) and Apo-lipoprotein Levels at Month 12
Description: Lipid (cholesterol) and apo-lipoprotein (A and B) are biomarkers of glucose metabolism in blood. The method used for analyzes was positron emission tomography (PET) using radiolabelled [18F] -fluoro-deoxy-glucose (FDG). Baseline measurement was performed on Day 1. Change from baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) and Month 12
Population: ITT population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Grams per Liter
  Apolipoprotein A: number analyzed (Participants) | 32 | 31
  Apolipoprotein A | -0.0478 (0.29284) | -0.2058 (0.27424)
  Apolipoprotein B: number analyzed (Participants) | 32 | 31
  Apolipoprotein B | -0.0191 (0.18714) | -0.0006 (0.25070)
  Cholesterol: number analyzed (Participants) | 32 | 30
  Cholesterol | -0.2556 (0.69756) | 0.1340 (1.09229)

17. Secondary Outcome: Change From Baseline in Inflammatory Biomarkers (CD40, C-reactive Protein [CRP] , Interleukin [ IL ]-6, and Tumor Necrosing Factor [TNF]-Alpha)
Description: The inflammatory biomarkers namely CD40, C-reactive protein (CRP) , interleukin (IL)-6, and tumor necrosing factor (TNF)-alpha) were analyzed. Baseline measurement was performed on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) and Month 12
Population: ITT population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per Liter
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 39
Nanograms per Liter
  CD40: number analyzed (Participants) | 31 | 30
  CD40 | -236.79 (2500.30) | 130.543 (2580.16)
  CRP: number analyzed (Participants) | 31 | 30
  CRP | 0.8161 (5.94099) | -1.4800 (4.63565)
  IL-6: number analyzed (Participants) | 31 | 30
  IL-6 | 6.3390 (22.5103) | 2.6370 (11.1159)
  TNF-alpha: number analyzed (Participants) | 28 | 27
  TNF-alpha | 16.7893 (53.0817) | 3.8407 (15.9970)

18. Secondary Outcome: Change From Baseline in Insulin Sensitivity Measured by Homeostasis Model Assessment of Insulin Resistance (HOMA IR)
Description: This is a measure of assessing insulin sensitivity. HOMA IR was calculated by multiplying fasting insulin by fasting plasma glucose and dividing the multiplied digit by 22.5. All samples were collected under fasting condition. Baseline measurement was performed on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) and Month 12
Population: ITT population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: HOMA IR score
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 31 | 31
HOMA IR score | -0.2703 (12.6037) | -5.9910 (9.79511)

19. Secondary Outcome: Number of Participants by Apo-lipoprotein -e (APOE Epsilon)-4 Allele Subtype
Description: Participants were categorized into two major types namely those with APOE4 genotype and without APOE4 genotype. Further, 6 subtypes/ alleles of APOE4 gene (as mentioned in the categories below) were analyzed. Participants were also classified as having 0 or 1 or 2 copies of this gene.
Time Frame: Up to 12 months
Population: PGx population included all ITT participants with evaluable PGx data (had consented to genotyping, provided and identified blood sample for genotyping and were successfully genotyped for at least one of the genetic markers under study). Only those participants available at time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 30 | 29
Participants
  With APOE4 gene | 24 | 15
  Without APOE4 gene | 6 | 14
  With E4E4 allele | 7 | 6
  With E3E4 allele | 17 | 8
  With E2E4 allele | 0 | 1
  With E3E3 allele | 5 | 12
  With E2E3 allele | 1 | 1
  With E2E2 allele | 0 | 1
  2 copies of APOE4 gene | 7 | 6
  1 copies of APOE4 gene | 17 | 9
  0 copies of APOE4 gene | 6 | 14

20. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Adverse event (AE) is an unfavorable change in the health of a participant, including abnormal laboratory findings, that happens during a clinical study or within a certain time period after the study has ended. This change may or may not be caused by the intervention being studied. Serious adverse event (SAE) is an adverse event that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect. Medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered serious adverse events if they put the participant in danger or require medical or surgical intervention to prevent one of the results listed above.
Time Frame: Up to 12 months
Population: All subjects population included all randomized subjects who receive at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 40 | 40
Participants
  Any AE | 32 | 33
  Any SAE | 6 | 4

21. Secondary Outcome: Number of Participants With Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Outside the Concern Range at Month 12
Description: Number of participants with SBP or DBP outside the defined range of clinical concern were collectively presented for any time on-treatment period. SBP of <90 millimeters of mercury (mmHg) and >140 mmHg was considered as of clinical concern. DBP of <50 and >90 mmHg was considered as of clinical concern. Increase in SBP from Baseline of >=40 mmHg and Decrease of >=30 mmHg was also recorded. Increase in DBP from Baseline of >=30 mmHg and Decrease of >=20 mmHg was also recorded.
Time Frame: At Month 12
Population: All subjects population. Only the participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 40
Participants
  SBP, >140 or <90 | 20 | 23
  SBP, Increase from Baseline>=40 | 1 | 3
  SBP, Decrease from Baseline>=30 | 12 | 13
  DBP, >90 or <50 | 5 | 2
  DBP, Increase from Baseline>=30 | 1 | 1
  DBP, Decrease from Baseline>=20 | 3 | 7

22. Secondary Outcome: Number of Participants With Heart Rate/ Pulse Rate Outside the Concern Range at Month 12
Description: Heart rate was measured in supine position. Number of participants with any time on-treatment values of heart rate values outside the clinical concern were presented. Heart rate values of >100 or <50 were considered as of clinical concern. Increase in heart rate from Baseline of >=30 beats per minute (bpm) and decrease in heart rate from Baseline of >=30 bpm was also recorded and presented.
Time Frame: At Month 12
Population: All subjects population. Only those participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Rosiglitazone: Eligible participants received unit oral dose of visually matching Placebo 4 mg for one month. Participants received escalated dose of 8 mg matching placebo for next 12 months and were followed-up to 30 days.
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 39 | 40
Participants
  Heart rate >100 or <50 | 4 | 3
  Increase in heart rate from Baseline of >=30 | 2 | 4
  Dncrease in heart rate from Baseline of >=30 | 0 | 0

23. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Parameters at Screening and Follow-up
Description: Two screening visits were arranged within 30 days of Day 1 of screening period and within 7 to 10 days of Day 1 of screening period. Follow-up period was arranged within 14 days of the last dose (post 12 months) of the study drug. Data for only the participants with abnormal ECG values has been presented.
Time Frame: At screening (within 1 month of Day 1) and follow-up period (within 2 weeks of final dose [12 months])
Population: All subjects population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 40 | 40
Participants
  At screening | 18 | 18
  At follow-up | 5 | 10

24. Secondary Outcome: Number of Participants With Body Weight and Height Outside the Clinical Concern at Month 12
Description: Body weight and height are the parameters of physical examination. Body weight is also a measure of fluid retention. Body weight increase or decrease of >= 7 % was considered as of clinical concern. Since there would be no or negligible (insignificant) change in height of a participant, no data has been presented for change from Baseline in height of participants after exposure to the study drug.
Time Frame: At Month 12
Population: All subjects population. Only those participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 33 | 31
Participants
  Increase from Baseline >=7% | 2 | 5
  Decrease from Baseline >=7% | 2 | 2

25. Secondary Outcome: Global and Regional CMRglu Index by APOE Epsilon-4 Allele Subtype at 12 Month
Description: The CMRglu was analyzed based on the APOE Epsilon-4 gene allele, whether it was present (positive) or was missing (negative) among the participants. The data has been presented for Month 12. Data has been presented for arithmetic mean; however, statistical analysis presented is based on LS means.
Time Frame: At Month 12
Population: PGx ITT population included all participants in ITT population who had evaluable PGx data (who consented to genotyping, provided an identified blood sample for genotyping and were successfully genotyped for at least one of the genetic markers under study. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: milligrams per cubic centimeter
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 40 | 40
milligrams per cubic centimeter
  Grey matter, APOE positive: number analyzed (Participants) | 16 | 11
  Grey matter, APOE positive | -0.2649 (0.58442) | -0.0903 (0.44270)
  Posterior cingulate gyrus, APOE positive: number analyzed (Participants) | 16 | 11
  Posterior cingulate gyrus, APOE positive | -0.2728 (0.69449) | -0.0987 (0.43553)
  Frontal lobe, APOE positive: number analyzed (Participants) | 16 | 11
  Frontal lobe, APOE positive | -0.2939 (0.66878) | -0.1046 (0.45385)
  Parietal lobe, APOE positive: number analyzed (Participants) | 16 | 11
  Parietal lobe, APOE positive | -0.2919 (0.60832) | -0.1404 (0.42635)
  Posterior temporal lobe, APOE positive: number analyzed (Participants) | 16 | 11
  Posterior temporal lobe, APOE positive | -0.2722 (0.48425) | -0.1175 (0.42617)
  Cerebellum, APOE positive: number analyzed (Participants) | 15 | 10
  Cerebellum, APOE positive | -0.2280 (0.54477) | -0.0375 (0.49150)
  Medial temporal lobe, APOE positive: number analyzed (Participants) | 16 | 11
  Medial temporal lobe, APOE positive | -0.1647 (0.39800) | -0.0004 (0.43929)
  Grey matter, APOE negative: number analyzed (Participants) | 3 | 12
  Grey matter, APOE negative | -0.1577 (0.06551) | -0.0107 (0.16654)
  Posterior cingulate gyrus, APOE negative: number analyzed (Participants) | 3 | 12
  Posterior cingulate gyrus, APOE negative | -0.2655 (0.11854) | 0.0141 (0.17927)
  Frontal lobe, APOE negative: number analyzed (Participants) | 3 | 12
  Frontal lobe, APOE negative | -0.1967 (0.09081) | -0.0323 (0.17438)
  Parietal lobe, APOE negative: number analyzed (Participants) | 3 | 12
  Parietal lobe, APOE negative | -0.1549 (0.08056) | -0.0362 (0.17425)
  Posterior temporal lobe, APOE negative: number analyzed (Participants) | 3 | 12
  Posterior temporal lobe, APOE negative | -0.1391 (0.11660) | -0.0443 (0.16786)
  Cerebellum, APOE negative: number analyzed (Participants) | 3 | 11
  Cerebellum, APOE negative | -0.1732 (0.05698) | 0.0742 (0.15230)
  Medial temporal lobe, APOE negative: number analyzed (Participants) | 3 | 12
  Medial temporal lobe, APOE negative | -0.1134 (0.06707) | 0.0026 (0.14382)
Statistical Analysis 1: Comparison: Placebo vs Rosiglitazone; For Grey matter, APOE Epsilon-4 status positive; Test type: Superiority or Other; p = 0.2800, Repeated measure mixed model; Mean Difference (Net) = 0.1154, 95% CI 2-sided [-0.0967 to 0.3275]
Statistical Analysis 2: Comparison: Placebo vs Rosiglitazone; For Grey matter, APOE Epsilon-4 status negative; Test type: Superiority or Other; p = 0.4159, Repeated measure mixed model; Mean Difference (Net) = 0.1337, 95% CI [-0.1931 to 0.4605]
Statistical Analysis 3: Comparison: Placebo vs Rosiglitazone; For posterior cingulate gyrus, APOE Epsilon-4 status positive; Test type: Superiority or Other; p = 0.2158, Repeated measure mixed model; Mean Difference (Net) = 0.1491, 95% CI 2-sided [-0.0897 to 0.3878]
Statistical Analysis 4: Comparison: Placebo vs Rosiglitazone; For posterior cingulate gyrus, APOE Epsilon-4 status negative; Test type: Superiority or Other; p = 0.2087, Repeated measure mixed model; Mean Difference (Net) = 0.2346, 95% CI 2-sided [-0.1350 to 0.6042]
Statistical Analysis 5: Comparison: Placebo vs Rosiglitazone; For Frontal lobe, APOE Epsilon-4 status positive; Test type: Superiority or Other; p = 0.3064, Repeated measure mixed model; Mean Difference (Net) = 0.1233, 95% CI 2-sided [-0.1162 to 0.3628]
Statistical Analysis 6: Comparison: Placebo vs Rosiglitazone; For Frontal lobe APOE Epsilon-4 status negative; Test type: Superiority or Other; p = 0.3500, Repeated measure mixed model; Mean Difference (Net) = 0.1734, 95% CI 2-sided [-0.1952 to 0.5420]
Statistical Analysis 7: Comparison: Placebo vs Rosiglitazone; For parietal lobe, APOE Epsilon-4 status positive; Test type: Superiority or Other; p = 0.2487, Repeated measure mixed model; Mean Difference (Net) = 0.1300, 95% CI 2-sided [-0.0937 to 0.3538]
Statistical Analysis 8: Comparison: Placebo vs Rosiglitazone; For parietal lobe, APOE Epsilon-4 status negative; Test type: Superiority or Other; p = 0.5521, Repeated measure mixed model; Mean Difference (Net) = 0.1038, 95% CI 2-sided [-0.2440 to 0.4516]
Statistical Analysis 9: Comparison: Placebo vs Rosiglitazone; For posterior temporal lobe, APOE Epsilon-4 status positive; Test type: Superiority or Other; p = 0.1760, Repeated measure mixed model; Mean Difference (Net) = 0.1384, 95% CI 2-sided [-0.0640 to 0.3409]
Statistical Analysis 10: Comparison: Placebo vs Rosiglitazone; For posterior temporal lobe, APOE Epsilon-4 status negative; Test type: Superiority or Other; p = 0.5952, Repeated measure mixed model; Mean Difference (Net) = 0.0837, 95% CI 2-sided [-0.2303 to 0.3978]
Statistical Analysis 11: Comparison: Placebo vs Rosiglitazone; For Cerebellum, APOE Epsilon-4 status positive; Test type: Superiority or Other; p = 0.4025, Repeated measure mixed model; Mean Difference (Net) = 0.0847, 95% CI 2-sided [-0.1169 to 0.2863]
Statistical Analysis 12: Comparison: Placebo vs Rosiglitazone; For Cerebellum, APOE Epsilon-4 status negative; Test type: Superiority or Other; p = 0.3081, Repeated measure mixed model95; Mean Difference (Net) = 0.1536, 95% CI 2-sided [-0.1458 to 0.4530]
Statistical Analysis 13: Comparison: Placebo vs Rosiglitazone; For medial temporal lobe, APOE Epsilon-4 status positive; Test type: Superiority or Other; p = 0.2964, Repeated measure mixed model; Mean Difference (Net) = 0.0839, 95% CI 2-sided [-0.0758 to 0.2436]
Statistical Analysis 14: Comparison: Placebo vs Rosiglitazone; For medial temporal lobe, APOE Epsilon-4 status negative; Test type: Superiority or Other; p = 0.2101, Repeated measure mixed model; Mean Difference (Net) = 0.1536, 95% CI 2-sided [-0.0892 to 0.3963]

26. Secondary Outcome: Number of Participants With Hematological Data of Potential Clinical Concern (PCC) at End of Treatment (Month 12)
Description: Participants were analyzed for any abnormality in basophils, eosinophils, hemoglobin, lymphocytes, monocytes, neutrophils, segmented neutrophils, platelets, red blood cells, and white blood cells with data outside the respective reference ranges. The values higher (H) or lower (L) than the reference range were analyzed at each month. The parameter has not been presented for participants who did not have any abnormality.
Time Frame: At Month 12
Population: All subjects population. Only the participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 40 | 40
Participants
  Hemoglobin, Month 12, L: number analyzed (Participants) | 31 | 29
  Hemoglobin, Month 12, L | 0 | 1
  Neutrophils, Month 12, L: number analyzed (Participants) | 31 | 29
  Neutrophils, Month 12, L | 0 | 1
  Platelets, Month 12, L: number analyzed (Participants) | 30 | 28
  Platelets, Month 12, L | 0 | 1
  White cells, Month 12, L: number analyzed (Participants) | 31 | 29
  White cells, Month 12, L | 1 | 1
  Lymphoctes percentage, Month 12, L: number analyzed (Participants) | 33 | 31
  Lymphoctes percentage, Month 12, L | 1 | 0

27. Secondary Outcome: Number of Participants With Clinical Chemistry Data of PCC at End of the Treatment (Month 12)
Description: Participants were analyzed for any abnormality in albumin, alanine aminotransferases, alkaline phosphatase, apolipoprotein A, apolipoprotein B, aspartate aminotransferases, Vitamin B12, direct bilirubin, indirect bilirubin, total bilirubin, cholesterol, creatinine, C-reactive protein, serum glucose, and non-fasting glucose, with data of PCC range. The values higher (H) or lower (L) than the reference range were analyzed at each month. The parameter has not been presented for participants who did not have any abnormality.
Time Frame: At Month 12
Population: All subjects population. Only the participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 40 | 40
Participants
  Direct bilirubin, H: number analyzed (Participants) | 34 | 31
  Direct bilirubin, H | 1 | 0
  Cholesterol, H: number analyzed (Participants) | 34 | 31
  Cholesterol, H | 1 | 0
  Glucose, H: number analyzed (Participants) | 32 | 31
  Glucose, H | 1 | 0
  Low density lipoprotein cholesterol, H: number analyzed (Participants) | 34 | 31
  Low density lipoprotein cholesterol, H | 2 | 5

ADVERSE EVENTS:
Time Frame: Up to 13 months
Description: All subjects population was used to report AEs and SAEs.
Arm/Group | Placebo | Rosiglitazone
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 6/40 | 4/40
Other Adverse Events (participants affected / at risk) | 32/40 | 33/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | Rosiglitazone (N=40)
LABYRINTHITIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
UROSEPSIS (Infections and infestations) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
FAECALOMA (Gastrointestinal disorders) | 0 | 1
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | Rosiglitazone (N=40)
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Dizziness (Nervous system disorders) | 3 | 3
Edema peripheral (General disorders) | 0 | 3
Herpes zoster (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Dementia Alzheimer's type (Nervous system disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 5 | 2
Fatigue (General disorders) | 1 | 2
Gait disturbance (General disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 2
Joint sprain (Injury, poisoning and procedural complications) | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Pneumonia (Infections and infestations) | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Agitation (Psychiatric disorders) | 2 | 0
Blood pressure increased (Investigations) | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Frequent bowel movements (Gastrointestinal disorders) | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.